CLINICAL TRIAL: NCT04348318
Title: Advance Directive Implementation and Scientific Evaluation (ADVISE) Study
Brief Title: Advance Directive Implementation and Scientific Evaluation Study
Acronym: ADVISE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00584; me20Sutter2
Record Dates: First submitted 2020-04-07; First posted 2020-04-16 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Loss of Capability of Judgement
Keywords: advance directives; life-sustaining treatment; neurocritical illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: health related personal data extraction from digital medical records — health related personal data extraction from digital medical records (i.e. patient characteristics; start, end and duration of hospitalization and ICU stay; admitted from another hospital, nursing home or comes with emergency medical Service; formal data of written advance directives; data of unwritten advance directive; information on the contents of the advance directives (regarding life-worthy conditions, health care agents, resuscitation, pain management, artificial nutrition, hydration, surgeries, renal replacement, mechanical circulation, mechanical ventilation, pacemaker, administration of blood products, treatment of infections, organ donation, autopsy); patient history; clinical data; therapeutic features; outcome at discharge; knowledge regarding relatives and their level of information about the advance directives; discussion of euthanasia and self-determination of dying.

SUMMARY:
This study is to better understand the use of advance directives, their implementation in the intensive care unit, and their effects on outcome. Data from the digital medical records of all consecutive adult patients admitted to the intensive care unit at the University Hospital Basel from 2011 to 2023 are retrospectively extracted. Descriptive analyses will be applied to report the proportion of patients with an advance directive. In-hospital outcome (defined as survival, Glasgow Outcome Score, and return of neurologic function to premorbid baseline) will be compared between patients with and without advanced directives

ELIGIBILITY:
Inclusion Criteria:

* adult patients treated for more than 48 hours in the intensive care unit (post-operative or internal medicine) of the University Hospital Basel in the years 2011-2023

Exclusion Criteria:

* Patients with documented refusal of the general consent.
* Patients who have been treated in the intensive care unit for less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all consecutive adult patients (i.e., ≥18 years of age) treated in the intensive care unit at the University Hospital Basel from 2011 to 2023.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
proportion of patients without predefined health care agents and/or completed advance directives | at baseline
  Descriptive analyses will be applied to report the proportion of patients with an advance directive. The core components of the advance directives will be analyzed regarding their translation into clinical practice. Patient and disease related characteristics will be compared between patients with and without advance directives applying the Chi-square and Fisher's exact test (where appropriate) for comparisons of proportions and the Mann-Whitney-U-test for the comparisons of continuous variables.
number of adequate translations of directives into clinical practice | at baseline
  Descriptive analyses will be applied to report the proportion of patients with an advance directive. The core components of the advance directives will be analyzed regarding their translation into clinical practice. Patient and disease related characteristics will be compared between patients with and without advance directives applying the Chi-square and Fisher's exact test (where appropriate) for comparisons of proportions and the Mann-Whitney-U-test for the comparisons of continuous variables.

SECONDARY OUTCOMES:
In-hospital outcome (defined as survival and return of neurologic function to premorbid baseline) | at baseline
  In-hospital outcome (defined as survival and return of neurologic function to premorbid baseline) will be compared between patients with and without advanced directives applying the Chi-square and Fisher's exact test (where appropriate) for comparisons of proportions and the Mann-Whitney-U-test for the comparisons of continuous variables.
In-hospital outcome (defined as Glasgow Outcome Score) | at baseline
  scale of patients with brain injuries that groups victims by the objective degree of recovery.The scale consists of five ordinal outcome categories: good recovery (able to live independently, able to return to work or school), moderate disability (able to live independently, unable to return to work or school), severe disability (able to follow commands, unable to live independently), persistent vegetative state (unable to interact with the environment, unresponsive), and death.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, PD Dr. med, Principal Investigator — Clinic for Intensive Care Medicine, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - Clinic for Intensive Care Medicine, University Hospital Basel, Basel

REFERENCES:
- [Derived] Baumann SM, Vock D, Kliem PSC, Amacher SA, Erne Y, Grzonka P, Berger S, Lohri M, Hunziker S, Gebhard CE, Nebiker M, Cioccari L, Sutter R. Prevalence, clinical impact and associated patient-centred outcomes of advance directives in Swiss intensive care units: Results from the retrospective ADVISE Study. Swiss Med Wkly. 2025 Sep 24;155:4625. doi: 10.57187/s.4625. PMID 41085533